CLINICAL TRIAL: NCT07301762
Title: Using Automated Manual Lymphatic Drainage Therapy to Optimize Glymphatic Function in Patients With Obstructive Sleep Apnea: Proof-of-Concept Open-Label Trial
Brief Title: Automated Manual Lymphatic Drainage Therapy to Improve Glymphatic Function in OSA Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Diego Zaquera Carvalho, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25-008009
Record Dates: First submitted 2025-12-21; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea (OSA); OSA; Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Other): Open-Label intervention
  Interventions: Device: Automated manual lymphatic drainage therapy (AMLDT) device

INTERVENTIONS:
Device: Automated manual lymphatic drainage therapy (AMLDT) device — The AMLDT device (Neuroglide) is an FDA-cleared Class II medical device (K202693) for over-the-counter use for pain. It mimics manual lymphatic drainage through a pneumatic mat that performs rhythmic inflation and deflation in ascending fashion.

SUMMARY:
The purpose of this research is to investigate whether enhancing systemic lymphatic drainage improves glymphatic function in patients with obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
This proof-of-concept, pre-post open-label clinical trial will enroll 12 adult patients aged 50 and older with previously treated OSA (≥6 months of CPAP adherence). Participants will undergo biomarker testing and sleep architecture analysis using ambulatory home sleep trackers (Somfit) before and after one month of nightly AMLDT intervention.

The significance of this study lies in its potential to uncover a novel, non-invasive therapeutic approach to enhance glymphatic clearance during sleep in OSA patients. The anticipated findings may inform future strategies for mitigating the risk of neurodegenerative diseases through targeted manipulation of the lymphatic system.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years and older
* Diagnosed with obstructive sleep apnea
* On stable, effective, and compliant CPAP therapy for a minimum of 6 months
* Willing and able to provide informed consent
* Willing and able to use automated manual lymphatic drainage device (Neuroglide) nightly for 1-month and participate in at-home sleep monitoring
* Stable on a medication regimen for comorbid medical or mental health disorders for at least 3 months and not planning to undergo therapy adjustment during trial

Exclusion Criteria:

* Chronic kidney disease (glomerular filtration rate (GFR) < 60 mL/min/1.73 m² for 3 months or more), due to its potential impact on serum biomarker clearance
* Other primary sleep disorders aside from OSA (i.e., narcolepsy, REM Sleep behavior disorder, chronic insomnia, restless legs syndrome), circadian rhythm disorder or shift work
* Chronic neurological disorders (e.g. Multiple sclerosis, epilepsy, neurodegenerative disorders, ALS), due to their impact on biomarkers. History of headache (<15 days a month) and stroke (over 6 months prior to enrollment) are allowed
* Physical limitations preventing the use of Neuroglide device (e.g. inability to lay on the back due to pain, inability to setup the device due to limb dysfunction/weakness)
* Physical limitations preventing the use or function of Somfit, including forehead skin lesions, history of adhesive allergies, implanted electronic devices (e.g. pacemakers) or the use of CPAP masks with forehead support/bar/pad (Fisher & Paykel Vitera, Fisher & Paykel Eson, ResMed Mirage Quattro, ResMed Ultra Mirage Full Face Mask, Philips Respironics ComfortGel Blue), because the forehead piece of the mask would prevent the appropriate application of Somfit for at-home sleep monitoring. Because Somfit algorithms are based on physiological signals that include heart rate and it has not been validated in patients with persistent arrhythmia, we will exclude patients with history of atrial fibrillation and high PVC burden to avoid inaccurate estimates.
* Acute cardiopulmonary disorders, infections, injury at/near the application site, abnormal lymphatic system due to previous surgery involving lymphatics or chronic lymphedema, acute inflammatory process (e.g. recent knee/hip surgery, upper respiratory tract infection, cancer not in remission)
* Kokmen short test of mental status < 34 (concern for mild cognitive impairment)
* Inability to comply with study procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Difference in serum biomarkers | Baseline and Day 31
  Samples will be processed and tested for:
  * Aβ42
  * Aβ40
  * Aβ42/Aβ40 ratio
  * Phospho-tau 217 (p-tau-217)
  * Neurofilament light chain (NfL)
  * Glial fibrillary acidic protein (GFAP)

SECONDARY OUTCOMES:
Differences in Pittsburgh Sleep Quality Index (PSQI) | Baseline and Day 31
  Differences in Pittsburgh Sleep Quality Index (PSQI) scores. Scoring ranges from 0-21 with higher scores indicating poorer sleep quality.

OTHER OUTCOMES:
Differences in sleep macro-structure and microstructure | Baseline and Day 31
  Assessment of correlation between changes in sleep macrostructure (Nonrapid eye movement sleep stages 1-3 [%], sleep duration [minutes], sleep efficiency [%]) and microstructure (power spectral density of slow wave activity [µV²/Hz]) and changes in serum biomarkers (1-42/1-40 [ratio], pTau181 [pg/mL], neurofilament light chain [pg/mL], and GFAP [pg/mL] ).

CONTACTS AND LOCATIONS:
Overall Officials: Diego Zaquera Carvalho, M.D., M.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No